CLINICAL TRIAL: NCT04810000
Title: The Effect of Releasing the Tourniquet in Total Knee Replacement Before Closure on the Blood Loss , Joint Effusion , Hematoma Formation and Wound Complication
Status: Completed | Type: Observational
Sponsor: Yazan Saleh Rajab Hammad (Other)
Responsible Party: Sponsor-Investigator, Yazan Saleh Rajab Hammad, Sponsor-Investigator - Senior orthopedic surgery resident, University of Jordan
Organization: University of Jordan (Other)
Other Study IDs: 10/2018/3489
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hematoma; Arthroplasty Complications
Keywords: Tourniquet; Intra articular Hematoma; Total Knee Replacement
MeSH Terms: conditions — Hematoma | interventions — Tourniquets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group A: Group A ( Tourniquet release before wound closure and hemostasis ensured )
  Interventions: Device: tourniquet
- Group B: Group B ( Tourniquet release after wound closure )
  Interventions: Device: tourniquet

INTERVENTIONS:
Device: tourniquet — Tourniquet release before/after wound closure

SUMMARY:
The study , observe the effect of releasing the Tourniquet in total knee replacement surgery before closure in comparison with releasing it after wound closure

The effect was assessed by Hb drop post operative and Hematoma formation ( measured by ultrasound ) as well as the wound complication

DETAILED DESCRIPTION:
The study is conducted in tertiary university hospital as a referral hospital for joint arthroplasty , the patients was informed about the study and consent was taken , the same operator , same theater and the same prosthesis company as well as the same radiologist during the study period.

the patient randomly assigned to either group A (Tourniquet release before closure of the wound and hemostasis ensured ) , or a group B ( Tourniquet release after wound closure )

post operative Hb drop was studied between the groups , and each patient underwent ultrasound measurement of the intraarticular hematoma . The wound complication between the groups was also studied .

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthrosis

Exclusion Criteria:

* Rheumatoid arthritis
* post traumatic arthritis
* revision knee replacement
* patients on anticoagulant/antiplatelet except acetylsalicylic acid 80-100 mg

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study was conducted in University hospital in the Capital city , the patients were from all around the country - Jordan - , as the hospital is as tertiary hospital most of the patients were above 60 , mostly female
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin(HG) drop | ( pre-operative and post-operative day 2)
  The difference in HG drop
Intra articular Hematoma formation | day three post operative hematoma formation
  the difference in Intra articular ( knee ) Hematoma collection between the groups on day 3 post operative

CONTACTS AND LOCATIONS:
Overall Officials: Yazan S Hammad, MD, Principal Investigator — Jordan University Hospital
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
the measurement of hemoglobin drop and intra articular hematoma measurement by ultrasound